CLINICAL TRIAL: NCT04741113
Title: The Effect of an Education Module to Reduce Weight Bias Among Healthcare Professionals in a Private Hospital Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Shiri Sherf Dagan, Dr. Shiri Sherf-Dagan, Dietitian and Epidemiologist, Assuta Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0008-20-ASMC
Record Dates: First submitted 2021-01-11; First posted 2021-02-05 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Obese, Stigma
MeSH Terms: conditions — Obesity; Social Stigma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group -educational module (Experimental): The study intervention will include an online 15-minute educational module with four sections: a) Knowledge about obesity; b) Weight bias definition and impact; c) Strategies to reduce weight bias; d) A short quiz.
  The module will be based on relevant literature and expert opinion. The module will be sent to participants via secured link.
  Interventions: Other: An online 15-minute educational module
- Control group (No Intervention): No intervention

INTERVENTIONS:
Other: An online 15-minute educational module — An online 15-minute educational module with four sections: a) Knowledge about obesity; b) Weight bias definition and impact; c) Strategies to reduce weight bias; d) A short quiz.
  The module will be based on relevant literature and expert opinion
  Arms: Intervention group -educational module

SUMMARY:
Although scientific bodies have recognized obesity as a disease, obese people are often stigmatized, facing discrimination, and accusations that they are responsible to their condition due to their lack of willpower by healthcare professionals. However, experimental research to reduce weight bias among healthcare professionals is lacking, and published studies to date are methodologically flawed, including lack of randomization, lack of control group and small sample size.

The study is designed to evaluate the effect of a comprehensive online education module on knowledge about obesity and weight bias in a convenience sample in a private hospital setting.

This is an interventional study conducted among all Assuta Medical Centers healthcare employees including physicians, bariatric surgeons, nurses, dietitians, social workers, physiotherapists, pharmacists, imaging department technicians, laboratory workers, patient services assistants and medical secretariats. Participants who will confirm their consent to participate in the study, will be randomized into two arms: intervention vs. control (with no intervention). The study intervention will include an online 15-minute educational module which will be based on relevant literature and expert opinion and will include four sections: a) Knowledge about obesity; b) Weight bias definition and impact; c) Strategies to reduce weight bias; d) A short quiz. At baseline, one week and one-month post intervention, both groups will respond to an anonymous on-line survey on knowledge about obesity and weight stigma. Moreover, data on demographic parameters of study participants will be collected.

ELIGIBILITY:
Inclusion Criteria:

* All Assuta Medical Centers healthcare employees will be recruited to the study

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Weight stigma | Change from Baseline at 1 month post intervantion
  Questionnaires on weight stigma

SECONDARY OUTCOMES:
Knowledge about obesity | Change from Baseline at 1 month post intervantion
  Questionnaire on knowledge about obesity

CONTACTS AND LOCATIONS:
Locations (1):
- Assuta Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sherf-Dagan S, Kessler Y, Mardy-Tilbor L, Raziel A, Sakran N, Boaz M, Kaufman-Shriqui V. The Effect of an Education Module to Reduce Weight Bias among Medical Centers Employees: A Randomized Controlled Trial. Obes Facts. 2022;15(3):384-394. doi: 10.1159/000521856. Epub 2022 Jan 21. PMID 35066508